CLINICAL TRIAL: NCT04476394
Title: A Single-center, Open, Single Dose Mass Balance Study to Assess the Absorption, Metabolism, Excretion of [14C]-20 mg/100 μCi Anaprazole Sodium Enteric-coated Capsule in Chinese Health Adult Male Subjects
Brief Title: Open-label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of a Single Oral Dose of [14C]-20 mg/100 μCi Anaprazole Sodium Enteric-coated Capsule in Healthy Adult Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3571-MB-1005
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-04

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Administered orally once
  Interventions: Drug: [14C]-Anaprazole Sodium enteric-coated capsule

INTERVENTIONS:
Drug: [14C]-Anaprazole Sodium enteric-coated capsule — [14C]-Anaprazole Sodium enteric-coated capsule

SUMMARY:
This is an open-label, single-dose, absorption, metabolism, excretion, and mass balance study following a single oral dose of [14C]-20 mg/100 μCi Anaprazole Sodium enteric-coated capsule in healthy adult male subjects. Whole blood, plasma samples will be collected at hour 0 pre-dose and 1，2，3，4，5，6，8，12，24，48，72，96，120，144，168 hours post-dose (tentative, adjusted according to plasma drug concentration); urine samples will be collected at hour 24 pre-dose and 0-4，4-8，8-12，12-24，24-48，48-72，72-96，96-120，120-144，144-168，168-192，192-216，216-240 hours post-dose (tentative, adjusted according to sample recovery rate) ; fecal samples will be collected at hour 24 pre-dose and 0-24，24-48，48-72，72-96，96-120，120-144，144-168，168-192，192-216，216-240 hours post-dose (tentative, adjusted according to sample recovery rate) following the start of administration to measure total radioactivity and plasma drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

* 1.The subject is a Chinese adult male, aged 18 to 45 years, inclusive.
* 2.The subject weighed at least 50.0 kg and had a body mass index (BMI) between 19.0 kg/m^2 and 26.0 kg/m^2, inclusive.
* 3. Participants with evaluations of vital signs, physicial examination results,clinical laboratory and ECG testing outside the reference range that are deemed not clinically significant at investigator discretion at screening.
* 4.The subject with childbearing potential agrees that the subject and his sexual partner use adequate contraception from signing of informed consent throughout the duration of the study and for 6 months after study completion.
* 5.The subject is capable of understanding and complying with protocol requirements, and signed and dated a written informed consent form voluntarily

Exclusion Criteria:

* 1.Has clinical significant drug allergy or allergic disease history(Such as asthma, urticaria, eczema dermatitis, etc), or has hypersensitivity or allergy to investigatory drugs or related supplements；
* 2.Has clinical significant ECG abnormal history or family history of long QT syndrome(Grandparents, parents and siblings)
* 3.Any disease or medical history that may significantly affect the absorption, distribution, metabolism, and excretion of drugs, or any condition that may pose a hazard to the subject. Such as:

  * Inflammatory bowel disease, gastric ulcer, duodenal ulcer, gastrointestinal / rectal bleeding, persistent nausea, or other clinically significant gastrointestinal abnormalities;
  * Has suffered from gastrointestinal diseases or complications that may affect the absorption of drugs (ie: malabsorption, gastroesophageal reflux, peptic ulcer, erosive esophagitis, frequent heartburn) within 6 months before screening or had history of gastrointestinal surgery (for example: gastrectomy, gastrointestinal anastomosis, intestinal resection, gastric bypass, gastric segmentation or gastric banding, cholecystectomy, except for appendicitis surgery and proctectomy);
  * Evidence of liver disease or clinically impaired liver function at the time of screening (eg AST, ALT or total bilirubin> 1.5 times ULN);
  * A history or evidence of nephropathy or renal insufficiency at the time of screening, showing clinically significant abnormality of creatinine or abnormal urine composition (such as proteinuria, creatinine> 176.8 umol / L, etc.)
  * Has difficulty swallowing oral preparations.
* 4.Thyroid stimulating hormone (TSH)> ULN; or serum free triiodothyronine (FT3)> ULN; or serum free thyroxine (FT4)> ULN at the time of screening;
* 5. Frequent smokers and alcoholics within 3 months before screening (smoke more than 5 cigarettes / day, drink more than 21 units of alcohol per week, 1 unit = 360 mL beer or 45 mL liquor or 150 mL wine), or can't stop using any tobacco products, and alcohol intake during the study period ; or those who have a positive alcohol breath test before enrollment;
* 6. Has received any investigational compound (including post-marketing investigational drugs) or participated in clinical trials of any drugs /devices within 3 months before screening;
* 7. A history of drug abuse within 12 months before screening or a positive urine test result at screening;
* 8. Has used any prescription drugs, non-prescription drugs (including chemical drugs, vitamin drugs, Chinese herbal medicines, etc.) within 4 weeks before administration of investigational drugs;
* 9. Has taken foods that affect CYP3A4 (such as grapefruit or beverages containing grapefruit) within 2 weeks before administration of investigational drugs;
* 10. Human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis C antibody, and Treponema pallidum specific antibody test results were positive at screening;
* 11. Has difficulty in venous blood collection or halo acupuncture;
* 12.Blood donation / blood loss ≥200 mL within 1 month, or ≥400 mL within 3 months before screening; or has blood donation plan during the period of medication of investigational drugs and within 3 months after drug withdrawal;
* 13. Has special dietary requirements and cannot follow the unified dietary arrangements;
* 14. Has particpated in another clinical study with radioactive labeling within 1 year before administration.
* 15. Has significant radiation exposure (Radiation exposure from chest X-ray, CT scan or barium meal examination more than once, or be engaged in radiation related occupations) within 1 year before administration.
* 16. Any conditions in which considered by investigator not be appropriate to participate in this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-08-03 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Cmax of Anaprazole according to total radioactivity concentration equivalents in whole blood and plasma | Hour 0 pre-dose and 1，2，3，4，5，6，8，12，24，48，72，96，120，144，168 hours post-dose (tentative, adjusted according to plasma drug concentration)
  Cmax is the peak plasma concentration
Tmax of Anaprazole according to total radioactivity concentration equivalents in whole blood and plasma | Hour 0 pre-dose and 1，2，3，4，5，6，8，12，24，48，72，96，120，144，168 hours post-dose (tentative, adjusted according to plasma drug concentration)
  Tmax is the time to maximum plasma concentration
AUC of Anaprazole according to total radioactivity concentration equivalents in whole blood and plasma | Hour 0 pre-dose and 1，2，3，4，5，6，8，12，24，48，72，96，120，144，168 hours post-dose (tentative, adjusted according to plasma drug concentration)
  AUC is area under the plasma concentration-time curve
Cumulative excretion and cumulative excretion rate in urine | Hour 24 pre-dose and 0-4，4-8，8-12，12-24，24-48，48-72，72-96，96-120，120-144，144-168，168-192，192-216，216-240 hours post-dose (tentative, adjusted according to sample recovery rate)
  Sum of the percent of the total radioactivity recovered in urine relative to the administered radioactivity dose
Cumulative excretion and cumulative excretion rate in feces | Hour 24 pre-dose and 0-24，24-48，48-72，72-96，96-120，120-144，144-168，168-192，192-216，216-240 hours post-dose (tentative, adjusted according to sample recovery rate)
  Sum of the percent of the total radioactivity recovered in feces relative to the administered radioactivity dose
Radioactivity spectrum indentification of metabolites in plasma | Hour 0 pre-dose and 1，2，3，4，5，6，8，12，24，48，72，96，120，144，168 hours post-dose (tentative, adjusted according to plasma drug concentration)
  plasma concentration of metabolites
Radioactivity spectrum indentification of metabolites in urine | Hour 24 pre-dose and 0-4，4-8，8-12，12-24，24-48，48-72，72-96，96-120，120-144，144-168，168-192，192-216，216-240 hours post-dose (tentative, adjusted according to sample recovery rate)
  Concentration of metabolites in urine
Concentration of metabolites in feces | Hour 24 pre-dose and 0-24，24-48，48-72，72-96，96-120，120-144，144-168，168-192，192-216，216-240 hours post-dose (tentative, adjusted according to sample recovery rate)
  Sum of the percent of the total radioactivity recovered in feces relative to the administered radioactivity dose